CLINICAL TRIAL: NCT02710409
Title: A Double-blind,Randomized,Positive-controlled, Non-inferiority Phase III Clinical Trial of An Inactivated Quadrivalent Influenza Vaccine (Split Virion) in Healthy Chinese Subjects Aged 3 Years and Older
Brief Title: A Phase III Clinical Trial of An Inactivated Quadrivalent Influenza Vaccine in Healthy Subjects Aged 3 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Jiangsu Jindike Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT031
Record Dates: First submitted 2016-03-12; First posted 2016-03-16 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Influenza
Keywords: safety, immunogenicity , quadrivalent influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Quadrivalent influenza vaccine (Experimental)
  Interventions: Biological: Quadrivalent influenza vaccine
- Trivalent influenza vaccine A (Active Comparator): Active Comparator A
  Interventions: Biological: Trivalent influenza vaccine A
- Trivalent influenza vaccine B (Active Comparator): Active Comparator B
  Interventions: Biological: Trivalent influenza vaccine B

INTERVENTIONS:
Biological: Quadrivalent influenza vaccine — 0.5 ml/vial, one dose, intramuscular injection on day 0
  Arms: Quadrivalent influenza vaccine
Biological: Trivalent influenza vaccine A — 0.5 ml/vial, one dose, intramuscular injection on day 0
  Arms: Trivalent influenza vaccine A
Biological: Trivalent influenza vaccine B — 0.5 ml/vial, one dose, intramuscular injection on day 0
  Arms: Trivalent influenza vaccine B

SUMMARY:
Influenza is an acute respiratory disease caused by influenza viruses. There are three types of the virus including A, B and C. Both type A and type B viruses can cause acute febrile respiratory tract infection, characterized by sudden fever, headache, muscle pain, cough, sore throat, nasal congestion and general malaise. The main transmission of influenza is through those highly contagious aerosol droplets containing influenza virus passed from infected people to susceptible population. Each year in the fall and winter infection of influenza is widespread in various age groups, with high incidence rate. Although influenza is generally a self-limiting disease, but in children, the elderly (especially those above 65 years old and those with chronic heart, lung, kidney, liver, blood or metabolic diseases such as diabetes or other certain diseases) and those with poor immunity function, influenza can easily lead to serious flu complications such as pneumonia, resulting in severe increase of morbidity and mortality.

In order to evaluate safety and immunogenicity of a quadrivalent influenza vaccine produced by Jiangsu Jindike Biotechnology Co., Ltd. a phase III clinical trial is planned to conduct in healthy Chinese subjects aged 3 years and older.

DETAILED DESCRIPTION:
Subjects will be randomized into three arms- Experimental Group, Active Comparator A and Active Comparator B by the ratio of 2:1:1.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 years and older
* Healthy subjects judged from medical history and clinical examination
* Subjects themselves or their guardians able to understand and sign the informed consent
* Subjects themselves or their guardians can and will comply with the requirements of the protocol
* Subjects with temperature <=37.0°C on axillary setting

Exclusion Criteria:

* Subject who has a medical or family history of any of the following: allergic history, seizure, epilepsy, brain or mental disease
* Any prior administration of influenza vaccine in last 6 month
* Subject who is allergic to any ingredient of the vaccine
* Female subject aged ≥18 years with a positive result after urine pregnancy test or during pregnancy or baby nursing period
* Subject with damaged or low immune function which has already been known
* Subject who had a seasonal influenza medical history in last 6 months
* Subject with acute febrile illness or infectious disease
* Major congenital defects or serious chronic illness, including perinatal brain damage
* Thrombocytopenia, blood coagulation disorder or bleeding difficulties with intramuscular injection
* Subject who has serious allergic history
* Subject with other medical history not suitable for vaccination such as fainting during injection
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of other research medicine/vaccine in last 30 days
* Any prior administration of any attenuated live vaccine in last 30 days
* Any prior administration of subunit or inactivated vaccines in last 14 days, such as pneumococcal vaccine
* Any medical, psychological, social or other condition judged by investigator, that may interfere subject's compliance with the protocol or signature on informed consent

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3664 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
the 95% confidence interval (CI) lower limit for the seroconversion against each corresponding flu strain after vaccination is≥40% in subjects aged 3-59 years and≥30% in subjects aged ≥60 years separately | 28 days after vaccination
  Immunogenicity outcomes were assessed in serum samples by Hemagglutination inhibition (HAI) assay. The lowest dilution used in the assay is 1/10. Seroconversion was defined as either a pre-vaccination HAI titer < 1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and ≥ four-fold increase in post-vaccination titer.
incidence of solicited adverse reactions after vaccination | 0-7 days after vaccination
  incidence of solicited adverse reactions (including systemic and local adverse reactions) after vaccination

SECONDARY OUTCOMES:
the 95% CI lower limit for the post-vaccination seroprotection rates against each corresponding flu strain is ≥70% | 28 days after vaccination
  A seroprotected subject is defined as a vaccinated subject with serum HAI titer≥ 1:40.
the post-vaccination mean geometric increases (GMIs) of HAI titer against each corresponding flu strain is≥2.5 in subjects aged 3-59 years and≥2.0 in subjects aged ≥60 years separately | 28 days after vaccination
  Hemagglutination inhibition (HI) titers were used to calculate post-vaccination mean geometric increases (GMIs) of each of the influenza vaccines.
incidence of unsolicited adverse reactions after vaccination | 0-28 days after vaccination
  incidence of unsolicited adverse reactions (including systemic and local adverse reactions) after vaccination
incidence of serious adverse event (SAE) after vaccination | 0-28 days after vaccination
incidence of serious adverse event (SAE) after vaccination | 29 days to 6 month after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Guanyun County Center for Disease Control and Prevention, Lianyungang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided